CLINICAL TRIAL: NCT03268395
Title: The Correlation of CO2 Measured by SenTec Transcutaneous Monitoring With Arterial Blood Gas CO2 Levels in Neonates
Brief Title: Correlation of CO2 Measured by Blood Gas vs Transcutaneous Monitor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memorial Health University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017.07.02
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Respiratory Complication
MeSH Terms: interventions — Blood Gas Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CO2 Measurement (Other): Each subject will received simultaneous arterial blood gas CO2 and transcutaneous CO2 monitor assessments. The correlation of these two measurements will be compared.
  Interventions: Diagnostic Test: Arterial Blood Gas and Transcutaneous CO2 Monitor

INTERVENTIONS:
Diagnostic Test: Arterial Blood Gas and Transcutaneous CO2 Monitor — Each patient will receive both an arterial blood gas and a transcutaneous CO2 monitor test.

SUMMARY:
The purpose of this clinical investigation is to compare transcutaneous CO2 (TCCO2) levels measured non-invasively using the SenTec Transcutaneous CO2 Monitor to PaCO2 levels measured on arterial blood gas (ABG) samples in neonatal patients being treated for respiratory distress in the Neonatal Intensive Care Unit (NICU) at Memorial University Medical Center.

DETAILED DESCRIPTION:
Background and Significance/Preliminary Studies Carbon dioxide (CO2) measurement is part of the fundamental respiratory evaluation in an ICU, as both high and low values of CO2 can have detrimental effects on neonatal health. The partial pressure of CO2 reflects ventilation, which is the elimination of carbon dioxide. The ABG sample is the clinical tool most commonly used to evaluate acid-base physiology at the bedside. It directly measures the pH, arterial partial pressure of oxygen, and arterial partial pressure of CO2. Though direct measurement of CO2 in the arterial blood is the most accurate way to assess the amount of CO2, it requires blood sampling from the arteries and does not provide continuous monitoring of CO2.

A non-invasive tool for measuring PaCO2, such as the SenTec monitor, can help decrease blood draws, thereby decreasing the incidence of iatrogenic anemia and the need for neonatal blood transfusions. Blood samples are collected through arterial lines, capillary heel sticks, or peripheral arterial punctures which are invasive and can be painful for the patient and may potentially result in injury. Although an ABG in neonates typically only requires 0.3mL-0.5mL of arterial blood, the need for frequent ABG sampling (every two to six hours) may result in a significant amount of iatrogenic blood loss. A newborn has a total blood volume of only 80mL/kg. In addition, the transcutaneous sensor has potential monitoring advantages as measurements are continuous rather than representative of a single point in time, as seen in ABGs. Continuous monitoring can help to avoid fluctuations in CO2 levels which can potentially result in neurologic injury in preterm babies, such as intraventricular hemorrhage and periventricular leukomalacia. One of the most beneficial aspects of the SenTec monitor is that it displays CO2 levels in real time, allowing clinicians to monitor trends and to intervene sooner if needed.

Previous studies have been conducted on transcutaneous monitors in newborns. One such study evaluated the CO-OXSYS Digital Sensor (also known as the V-Sign Digital Sensor) made by SenTec. 25 patients between the ages of 10 months to 79 years of age were studied. Each sensor was placed on the tragus of each patient's ear. An ABG was obtained fifteen minutes after sensor application and TCCO2 measurements were recorded at the same time. ABG samples were analyzed with a Rapidpoint 405 analyzer. A reliable correlation was found between the TCCO2 and the PaCO2 readings (R2-0.61, p=<0.001). It was noted that age and temperature did not affect the accuracy of the CO2 readings. This study concluded that with more sampling, the CO-OXSYS Digital Sensor would be useful in a variety of clinical settings.

A second study was performed assessing the SenTec monitor during neonatal High Frequency Oscillatory Ventilation. Fourteen neonatal patients were studied. The digital sensor was applied to each patient on varying body parts that included the left chest, right chest, and liver. Fifteen minutes after sensor application, an ABG was obtained and the simultaneously displayed TCCO2 measurement was recorded. ABG measurements were subsequently analyzed using a Siemens Rapidpoint 405 analyzer. A clinically acceptable correlation was found between the TCCO2 and PaCO2 readings (R2=0.807, p=<0.001). This study suggested the monitor could certainly be used as an alternative to ABGs.

In 2004 a study reviewed the TOSCA monitor, made by Linde Medical Sensors, which combined pulse oximetry and TCCO2 monitoring. This machine used a single ear sensor which worked at 42 degrees C to enhance blood flow in capillaries below the sensor. This study included 60 neonates who had an ear sensor placed on the right earlobe. Ten minutes after placement, an ABG was performed and compared to the TCCO2 reading. The transcutaneous readings were found to be clinically acceptable when compared to the ABGs. A secondary benefit of the transcutaneous monitoring on the earlobe was a decrease in the head movement of the neonate to aid in maintaining a patent airway. In addition, the sensor did not have to be removed for chest radiographs or while the parent was bonding with his or her infant in their lap (also known as "kangaroo care").

A recently completed study used the actual SenTec monitor I will be using. A total of 15 patients were included in this study with the following inclusion criteria:

Current weight > =1000grams Need for mechanical ventilation Arterial access Signed informed consent by parents/legal guardians The sensor was placed on the abdominal wall and when a routine ABG sample was obtained, the reading from the transcutaneous device was recorded. Photographs were also taken throughout the study to evaluate any injury to the skin from the monitor. The photographs were randomized and a blinded reviewer rated the photographs as normal, mild erythema, or burn/blistering. The reviewer of the photographs confirmed that there were no adverse skin changes. It was concluded that the TCCO2 measurements obtained correlated with the PaCO2 values.

Study Aims This research study is designed to assess the accuracy of SenTec transcutaneous monitors for CO2 monitoring in neonatal patients. The data from this research may be used to implement the SenTec monitors as part of the regular monitoring equipment used in the NICU at Memorial University Medical Center. These results will contribute to my course of study by aiding in my future research paper publication and poster presentation (to other ICU attendings).

Administrative Organization The Level III NICU at Memorial University Medical Center will be the sole participating unit. Registered nurses and/or respiratory therapists within the NICU will be collecting the routine ABG samples. Respiratory therapists within the NICU will analyze the ABG samples.

Study Design The design of the study will be an open-label, correlational prospective study. The study population will be any neonate weighing greater than one kg at birth requiring an arterial catheter for monitoring for cardiorespiratory distress. At the end of my study, if it is found that the SenTec digital monitor is as accurate and valid as the ABG samples collected and that no adverse skin changes are observed, I hope that the SenTec monitoring system will be implemented into Memorial's regular NICU monitoring equipment. With approval from the SenTec manufacturer, I will aim to write a paper and submit it to an appropriate neonatal or critical care journal for future publication. In addition to the paper, I plan to create a poster for presentation to critical care (PICU and NICU) unit staff (physicians, RTs, RNs, and NPs) at Memorial University Medical Center.

Study Procedures The sampling plan will include any neonate with a birth weight over 1000g, requiring an arterial line. Patients with significant pre-existing skin breakdown over the abdominal area will be excluded from the study. Recruitment will occur exclusively in the NICU. Consent will be obtained in the NICU once the arterial line has been placed. As the Principal Investigator, I, and/or other Dr. Daniel Sandler will obtain consent. We will provide the patient's parents with a summary of the protocol of the study and brochures providing information about the sensor and its manufacturer.

There will be no placebo study agents. This is going to be a validation study. The sensor will be stored in the NICU. The sensor will be placed on the patient by the patient's bedside RN. Potential adverse effects should be minor and limited to mild, local skin reactions.

Serial TCCO2 measurements will be compared to PaCO2 levels measured on arterial blood gas (ABG) samples obtained simultaneously on these patients. The sensor will be calibrated and applied to the skin according to manufacturer instructions. Whenever an arterial blood gas is collected for clinical indications, the transcutaneous monitor's reading will be simultaneously recorded in a data log including the patient's initial diagnosis, gestational age, sex, sensor location, birth weight, and body temperature. The skin of each infant will be closely inspected for injury (such as irritation or breakdown) before the skin probe is applied, and after each time that the probe is removed. Application skin sites will also be photographed on entry to and exit from the study, and whenever the probe is removed.

The photographs taken and the data log will be stored in an Excel document on a Memorial University Medical Center computer in the NICU. All study information will be password protected. Only the investigators (Charli Cohen, Dr. Daniel Sandler), and Eric Clayton, the study statistician, will have access to the study data collected.

Safety Monitoring Plan There is a slight risk for minor skin reactions from the probe. This sensor has been tested in newborns and it seems that any adverse skin events have been minimal. The probe has not yet been tested in extremely premature babies (weighing less than one kilogram at birth). We will constantly be monitoring the patient's safety during routine unit checks. The study investigators, with the assistance of NICU staff members, will identify, document, and report adverse events. A patient will be removed from the study if the skin reaction becomes severe. To carefully monitor for skin changes, photographs will be taken before and after application of the probe.

Analysis Plan

Hypotheses:

H0: Observed mean difference between PaCO2 and TCCO2 < 10 mmHg. Ha: Observed mean difference between PaCO2 and TCCO2 > 10 mmHg.

The study data will be analyzed using the Bland Altman technique for assessing agreement between two methods of clinical measurement6. Consistency between the PaCO2 and TCCO2 methods will be quantified by constructing limits of agreement (LoA). These limits are determined by using the observed mean and standard deviations of the differences between the two methods. A scatterplot will be constructed in which the Y-axis contains the differences in the paired measurements for each case (TCCO2 - PaCO2) and the X-axis contains the means of the same paired measurements ((TCCO2 + PaCO2)/2). A line representing the observed mean difference will be constructed parallel to the X-axis, as will two more lines at the points ± 1.96SD of the mean difference. These lines represent the LoA. 95% confidence intervals for the upper and lower LoA will be calculated. The pre-defined maximum acceptable difference between the methods of measurement has been determined as 10 mmHg. If the upper 95% confidence interval of the upper LoA and the lower 95% confidence interval of the lower LoA are both less than 10 mmHg from the observed mean difference, the H_0 will be accepted and the two measurement methods will be said to be in agreement.

Sample Size:

Using the published data and sample size methods, with α=0.05, β=0.20, expected mean difference (D = -3.21 mmHg), expected standard deviation (SD = 3.01 mmHg), and the clinically significant maximum allowed difference between the methods (δ=10 mmHg), the required minimum number of paired measurements is 266.

ELIGIBILITY:
Inclusion Criteria:

* Neonates in NICU with an arterial line

Exclusion Criteria:

* Birth Weight < 1000g

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-08-29 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Observed mean CO2 difference | 1 Minute
  The observed difference between arterial blood gas and transcutaneous CO2 monitor readings

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial University Medical Center, Savannah, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bernet-Buettiker V, Ugarte MJ, Frey B, Hug MI, Baenziger O, Weiss M. Evaluation of a new combined transcutaneous measurement of PCO2/pulse oximetry oxygen saturation ear sensor in newborn patients. Pediatrics. 2005 Jan;115(1):e64-8. doi: 10.1542/peds.2004-0946. Epub 2004 Dec 15. PMID 15601814